CLINICAL TRIAL: NCT03587064
Title: Non-inferiority Randomized Clinical Investigation of CRT-DX Versus CRT-D Systems
Brief Title: Comparison of CRT-D and CRT-DX Systems (CRT-NEXT)
Acronym: CRT-NEXT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associazione Portatori Dispositivi Impiantabili Cardiaci (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APDIC
Record Dates: First submitted 2018-06-14; First posted 2018-07-16 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure; Cardiac Resynchronization Therapy
Keywords: CRT-D; CRT-DX; Atrial pacing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-lead CRT implantation (CRT-D) (Active Comparator): In the 3-lead CRT implantation (CRT-D) group, conventional 3-lead CRT defibrillator system implantation will be performed. The CRT-D system is composed by three leads, one in atrium and two in both ventricles
  Interventions: Device: Conventional 3-lead CRT defibrillator system implantation
- 2-lead CRT implantation (CRT-DX) (Experimental): In the 2-lead CRT implantation (CRT-DX) group, 2-lead CRT defibrillator system implantation will be performed. The CRT-DX system is composed by two ventricular leads, the right one is provided with a dipole for atrial sensing
  Interventions: Device: 2-lead CRT defibrillator system implantation

INTERVENTIONS:
Device: Conventional 3-lead CRT defibrillator system implantation — Conventional 3-lead(1 atrial and 2 ventricular leads) system implantation
  Arms: 3-lead CRT implantation (CRT-D)
Device: 2-lead CRT defibrillator system implantation — 2-lead (2 ventricular leads with dipole for atrial sensing) DX system implantation
  Arms: 2-lead CRT implantation (CRT-DX)

SUMMARY:
The principal objective is to test non-inferiority of the CRT-DX system as compared to a conventional CRT-D system, in terms of the combined endpoint of mortality, hospitalizations due cardiovascular causes, any complication leading to loss of lead functionality, in the subset of patients without evidence of sinus dysfunction on optimal therapy.

DETAILED DESCRIPTION:
Resting heart rate is strongly associated with incident worsening Heart Failure (HF) and mortality. Current devices for cardiac resynchronization (CRT-D) normally provide atrio-ventricular (AV) sequential pacing modes during resynchronization, but the best pacing programming strategy is not clear.

On the one hand a basic rate of 50 to 70 bpm (optionally with some rate-responsive function) could be considered for therapy up-titration, specifically betablockers; on the other hand, increasing pacing rates may partially reduce benefits from resynchronization, reducing filling time and contractility reservoir.

The Pegasus investigation is the only large randomized investigation comparing DDD with 70 bpm basic rate to DDD(R) @40 bpm. Results showed no difference in investigation endpoints, including mortality and HF-hospitalization.

These results may support the use of a device implementing both a CRT function and a right ventricular single-lead with and an atrial sensing dipole (CRT-DX system). This system can track ventricular pacing and resynchronization following atrial sensing, even if it cannot provide atrial pacing support. It should be assessed whether such limitation is counterbalanced by the advantages related to the reduced number of necessary leads, with simplified implantation and less complications.

The objective of the investigation is to assess whether atrial pacing support is really necessary in the subset of patients with indication to CRT-D and no evidence of sinus dysfunction on optimal therapy. The investigation will test the hypothesis that a CRT-DX system is not inferior to a conventional CRT-D system in this class of subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥ 18 years old
2. Patients willing to participate in the investigation and signing the Patient Informed Consent (PIC) Form;
3. Indication to CRT-D implant according to current ESC Guidelines on cardiac pacing and cardiac resynchronization therapy
4. Sinus rhythm at time of implant;
5. Optimized medical therapy according to current ESC Guidelines
6. Rest heart rate (HR) >45 bpm at baseline ECG, with betablocker therapy at optimal medical dosage; or, if rest HR<45 bpm: maximum heart rate at the 6- minute walking test >85 bpm.

Exclusion Criteria:

1. Any indication to atrial pacing according to current guidelines;
2. Both: resting heart rate <45 bpm at baseline ECG, with betablocker therapy at optimal medical dosage and maximum heart rate at the 6-minute walking test <85 bpm;
3. NYHA Class IV;
4. Permanent Atrial Fibrillation
5. Replacement of/upgrading from previously implanted pacing system;
6. Dialysis patients;
7. Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint of Mortality, hospitalization due to cardiac causes and lead-related complications | 1 year
  It includes number of patients who experienced death, hospitalization due to cardiac causes, or any lead-related complication leading to loss of functionality (including lead dislodgement, conduction or insulation failure, loss of sensing or capture that couldn't resolved by reprogramming)

SECONDARY OUTCOMES:
Rate of implant revisions | 1 year
  Rate of implant revisions to add, replace, reposition, and remove an atrial pacing lead.
Rate of inappropriate therapy of the device | 1 year
  Inappropriate detections and interventions of high rate ventricular episodes.
Atrial pacing percentage | 1 year
  In the conventional CRT-D group, atrial pacing percentage.
Exercise test | 1 year
  Six minute walking test distance at one year
Device detected AT | 1 year
  Incidence of atrial tachyarrhythmias (AT)
Incidence of appropriate Ventricular therapy | 1 year
  Incidence of Ventricular Arrhythmias (VA) requiring therapy delivery
Incidence of events due to short-long-short sequence | 1 year
  Incidence of both VA and AT due to bradycardia or short-long-short sequence
Implant failure | 1 year
  Impossibility to implant any component (leads and device) of the initially planned system
Procedure times | 1 year
  Skin-to-skin and fluoroscopy time
Atrial sensing amplitude measured by device | 1 year
  Atrial sensing amplitude measured by devices in both investigation arms
Far field oversensing incidence | 1 year
  Incidence of far field oversensing episodes in both investigation arms

CONTACTS AND LOCATIONS:
Locations (24):
- Italy (24):
  - ASST Rhodense, Rho, Milano
  - Ospedale di Camposampiero, Camposampiero, Padova
  - AOU Ospedali Riuniti Ancona, Ancona
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S.Orsola Malpighi, Bologna
  - Fondazione Giovanni Paolo II, Campobasso
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele - Presidio Ferrarotto, Catania
  - Clinica Sant'Anna, Catanzaro
  - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro
  - Arcispedale Sant'Anna, Ferrara
  - Ospedale Santa Maria Nuova, Florence
  - Ospedale di Gorizia, Gorizia
  - Ospedale Vito Fazzi, Lecce
  - Ospedale Mater Salutis di Legnago, Legnago
  - Ospedale Carlo Poma, Mantova
  - IRCSS - Centro Neurolesi Bonino Pulejo, Messina
  - Ospedale San Gerardo, Monza
  - AOU Vanvitelli - Monaldi, Napoli
  - AO dei Colli - PO Monaldi, Napoli
  - Ospedale Federico II, Napoli
  - Azienda Ospedaliero - Universitaria di Parma, Parma
  - Fondazione Toscana Gabriele Monasterio, Pisa
  - Ospedale Giovanni Paolo II, Ragusa
  - Ospedale Molinette, Torino
  - Ospedali Riuniti Trieste, Trieste

IPD SHARING:
Plan to Share IPD: No